CLINICAL TRIAL: NCT06186570
Title: Efficacy of an Online-Based Self-Help Intervention for Auditory Hallucinations in Persons With Psychotic Disorders (ECHION)
Brief Title: Efficacy of an Online-Based Self-Help Intervention for Auditory Hallucinations in Persons With Psychotic Disorders
Acronym: ECHION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Kerem Böge, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECHION2024
Record Dates: First submitted 2023-12-05; First posted 2024-01-02 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Psychotic Disorders
Keywords: psychotic disorders; auditory hallucinations; voices; psychotherapy; self-help
MeSH Terms: conditions — Psychotic Disorders; Hallucinations

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with a parallel group design is used. The intervention group will receive the online-based self-help intervention immediately after the baseline assessment (T0), while the waitlist-control group will receive the online-based self-help intervention after study completion at T1. Both study conditions are allowed to continue standard scheduled treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online-Based Self-Help Intervention (Experimental): The online-based self-help intervention is implemented as a six-week self-help intervention that is primarily based on Metacognitive Training (MKT), Mindfulness-Based Group Therapy (MBGT), and elements of cognitive behavioural therapy. It is conducted online and includes worksheets, audio, and interactive files. Participants work themselves through the intervention, based on their own needs and speed. All participants are allowed to continue parallel implemented standard scheduled treatment (TAU; for a description of TAU, see the section below).
  Interventions: Behavioral: Online-Based Self-Help Intervention
- Waitlist-Control Group (No Intervention): The waitlist control group will not receive any additional intervention but is allowed to continue standard scheduled treatment (WL-TAU). This includes various forms of psychotherapeutic, pharmacologic, psychosocial, online, and other self-help interventions, either carried out individually or within a group. After study completion, participants in the waitlist-control group will equally receive the online-based self-help intervention.

INTERVENTIONS:
Behavioral: Online-Based Self-Help Intervention — See the description above.
  Arms: Online-Based Self-Help Intervention

SUMMARY:
The proposed clinical trial aims to examine the efficacy of an online-based self-help intervention for auditory hallucinations in persons with psychotic disorders. The intervention is primarily based on Metacognitive Training (MKT) and Mindfulness-Based Group Therapy (MBGT). The investigators will utilize a mixed-method study design within a randomized controlled trial. The intervention group will be compared with a waitlist-control group (WL-TAU). Both study conditions are allowed to continue standard scheduled treatment. The aim is to analyze the efficacy of and the subjective satisfaction with the intervention, based on self-report assessments evaluated from baseline (T0) to post-intervention after 6 weeks (T1).

DETAILED DESCRIPTION:
The investigators will identify eligible participants at various outpatient departments, suitable support groups, online platforms, and social media. An eligibility screening (in person or by telephone) to ensure the inclusion criteria and to introduce the study is held by the study assistant. All participants must sign an informed electronic consent after written and verbal study clarification. If persons are eligible for participation, they will be randomized according to a randomization plan by the electronic database RedCap. Due to the psychotherapeutic nature of the study, there will be no blinding. Participants in both study conditions will carry out self-reported measurements (online) at baseline (T0) and after the intervention phase of 6 weeks (T1). With an anticipated n = 25 of persons from the intervention group, there will be additionally conducted semi-structured interviews at T1 that aim to examine specific patterns of auditory hallucinations and satisfaction with the intervention. The final sample of the qualitative research part will be determined according to the principle of saturation (content-related). The data management plan includes standard procedures for data-handling such as using anonymized identification codes for patient data. Besides, the participants have the right to access their data, and the right to claim an annihilation. The data is being saved in an online database, only allowing researchers involved in the study to access the data.

ELIGIBILITY:
Inclusion Criteria:

* current experience of auditory hallucinations that appear at least once a week (measured over the PSYRATS).
* diagnosis of a schizophrenia-spectrum disorder according to the Diagnostical and Statistical Manual (5th edition) and/or the International Statistical Classification of Diseases and Related Health Problems (ICD-10), code F2x.x. In case of a suspected diagnosis or missing clinical diagnostic, we will apply the Mini-International Neuropsychiatric Interview (M.I.N.I.).
* stable psychiatric medication over at least one month, slight changes of dosage are allowed and will be evaluated by a trained psychiatrist.
* ability to give informed consent.
* willingness and ability to engage in the psychotherapeutic self-help intervention.
* availability of a mobile device and internet access.

Exclusion Criteria:

* neurological disorders that may affect cognitive functioning and condition after severe traumatic brain injury.
* acute suicidality, assessed at the previous screening procedures.
* auditory hallucinations in the context of other primary diagnoses e.g., post-traumatic stress disorder or borderline personality disorder.
* acute substance abuse other than nicotine and prescribed medication.
* current electroconvulsive therapy.
* current inpatient or day-care treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Frequency and distress of auditory hallucinations, PSYRATS | At baseline and post-intervention at week 6 (T1).
  The frequency and distress of auditory hallucinations measured by the hallucination subscale of the Psychotic Symptom Rating Scales (PSYRATS). Comparison between the intervention and control group, considering changes from baseline to post-intervention.

SECONDARY OUTCOMES:
Beliefs about voices, BAVQ-R | At baseline (T0) and post-intervention at week 6 (T1).
  Revised Beliefs About Voices Questionnaire (BAVQ-R), 35 items on a scale from 0 (disagree) to 3 (agree), including 5 subscales.
Hallucinatory experiences, LSHS-R | At baseline (T0) and post-intervention at week 6 (T1).
  Launay-Slade Hallucination Scale (LSHS-R), 12 items on a scale from 0 (certainly does not apply to me) to 4 (certainly applies to me).
Negative Symptoms, SNS | At baseline (T0) and post-intervention at week 6 (T1).
  Self-assessment of Negative Symptoms (SNS), 20 items on a scale from 0 (strongly disagree) to 2 (strongly agree).
Positive and Negative Affect, PANAS | At baseline (T0) and post-intervention at week 6 (T1).
  Positive and Negative Affect Schedule (PANAS), 20 items on a scale from 1 (not at all) to 5 (extremely).
Characteristics of Voices, Thinking Scale | At baseline (T0) and post-intervention at week 6 (T1).
  Thinking Scale (Moritz & Larøi, 2008), with 4 items addressing prevalent characteristics of voices (resemblances between imagined and real voices):
  1. "Loudness", using the following scale: 1 = "The voices are as loud as real voices", 2 = "The voices are louder than real voices", 3 = "The voices are lower than real voices", 4 = "The voices are actually audible".
  2. "Ego-Stability", using the following scale: 1 = "The voices reflect my own inner self", 2 = "The voices are saying things I would never think of or feel this way", 3 = "The voices can be influenced just as little as real voices".
  3. "Reality", using the following scale: 1 = "The voices are not particularly real", 2 = "The voices are nearly real", 3 = "The voices are absolutely indistinguishable from real voices".
  4. "Under which circumstances do the voices occur?", free-text answer.
Patient Satisfaction, ZUF-8 | At post-intervention at week 6 (T1) and only in the intervention group.
  Patient Satisfaction Questionnaire (ZUF-8), 8 items on a 4-point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No